CLINICAL TRIAL: NCT03834207
Title: A Federated Collaborative Care Cure Cloud Architecture for Addressing the Needs of Multi-morbidity and Managing Poly-pharmacy
Brief Title: A Study of the Usefulness & Usability of a Healthcare IT System for Managing Multi-morbidity and Poly-pharmacy
Acronym: C3-Cloud
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Christopher Marguerie (Other)
Collaborators: University of Warwick (Other); Biosistemak Institute for Health Systems Research (Other); Medixine (Unknown); SRDC (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Eurorec (Unknown); Empirica (Unknown); Örebro University, Sweden (Other); Osakidetza (Other); Region Jämtland Härjedalen (Other); Cambio Healthcare (Unknown)
Responsible Party: Sponsor-Investigator, Dr Christopher Marguerie, Consultant Rheumatologist/Associate Medical Director for Research, South Warwickshire NHS Foundation Trust
Organization: South Warwickshire NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 689181
Record Dates: First submitted 2019-01-02; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Type 2; Renal Failure; Heart Failure; Depression; Chronic Disease; Aging
Keywords: C3-Cloud; Multimorbidity; Diabetes Type 2; Heart Failure; Cardiac Failure; Depression; Renal Failure; Kidney Failure; Ageing; Computer System; Information Technology; Patient Empowerment; Guideline Reconciliation; Polypharmacy; Integrated Care; Clinical Decision Support
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency; Heart Failure; Depression; Chronic Disease; Patient Participation

STUDY DESIGN:
Intervention Model Description: A single intervention group that will use and evaluate the C3-Cloud system during the 12 month study. Please note that an anonymous group of patients meeting the same criteria will be identified retrospectively at the end of the study so that healthcare resource utilisation during the same period can be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Use of the C3-Cloud IT system
  Interventions: Device: Use of the C3-Cloud IT system

INTERVENTIONS:
Device: Use of the C3-Cloud IT system — Patients who are recruited to the intervention arm will use the C3-Cloud system during the pilot study.

SUMMARY:
To assess the acceptability of a personalised ICT tool that facilitates coordinated care planning, treatment optimisation and patient self-management for patients with multiple long term conditions and their team of health professionals.

DETAILED DESCRIPTION:
C3-CLOUD is a 4 year research project (information technology trial) funded by the EC to develop, pilot & evaluate a new clinical IT system to improve the management of elderly patients with multi-morbidity & poly-pharmacy. It will optimise patient education & self-management and foster closer collaborative working and shared decision making between healthcare professionals & patients using electronic multi-disciplinary care plans.

The main research question is - "Is the use of a personalised ICT tool that facilitates coordinated care planning, treatment optimisation and patient self-management acceptable to patients with multiple long term conditions and their team of health professionals?".

The 1st phase has focused on the development & testing of the system. The 2nd phase will involve a 12 month pilot (Feb 17-Jan 18) with max 602 patients (+/- the support of their informal care givers), and a minimum of 62 healthcare professionals in 3 European pilot sites in the UK, Sweden & Spain. An evaluation will be conducted using healthcare/treatment data & the completion of questionnaires by the study participants.

The C3-Cloud project structure is as follows:- Funded by the EC; Co-ordinated by Warwick University; 12 European partners involved, supplying technical, clinical & research expertise. These partners are based in the UK, Spain, Sweden, France, Turkey, Finland & Germany; and 3 European pilot sites involved in the study - Basque Country in Spain, Region Jamtland in Sweden and South Warwickshire in the UK.

The C3-CLOUD system consists of the following 2 integrated components. (i) C3DP - this component will be used by healthcare professionals in all 3 pilot sites to manage the care of the study patients. This system records e.g. patient identifiers, contact information, diagnoses, medication, treatments, encounters, risk factors, goals & activities for the patients etc. It also provides professionals with a clinical decision support module. (ii) a Patient Empowerment Platform (PEP) - used by patients (& carers where applicable) so that they can view & update their care plan. Patients can record information about themselves, their condition and their care, can view training materials & upload readings such as blood pressure etc. PEP also automatically takes information from the C3DP system above.

The study is aiming to recruit a minimum of 602 patients to the C3-CLOUD pilot study across all 3 pilot sites. Informed consent to participate in the study will be obtained. The patients must be aged 55+ and have at least 2 or more of the following chronic diseases - diabetes type 2, mild to moderate heart failure, moderate kidney failure and mild to moderate depression. They must also have a sufficiently high level of IT understanding and access to a suitable device/the internet, or must nominate a carer, family member or friend who does.

The patients who are recruited will receive care and treatment using the C3-CLOUD system and will have identifiable data collected about them by healthcare professionals in C3DP, and will use, and provide information about themselves, in the PEP system.

A separate cohort of max 602 patients will be identified retrospectively from local health records at the end of the study to create a 'control' group. These patients will match the same inclusion criteria. However, this control group will have no active role in the study and only their anonymised data will be utilised so that resource utilisation, medication use etc, can be compared for the two groups over the same period.

In the UK, the system will be used by a cross-section of healthcare professionals (minimum 62) across the 3 pilot sites. These will be the healthcare professionals who are most likely to be involved ordinarily in treating the patients during the study.

In addition to the clinical data captured above, the intervention group patients, their carers and the healthcare professionals involved in the project will participate in a series of system/project evaluations before, during and after the study. This will be done through anonymised questionnaires.

Healthcare utilisation & outcome data will be collected about intervention AND control group patients from local health records systems in an anonymised format. Evaluation data for the intervention group patients will also be extracted from the C3-Cloud system itself in an anonymised format.

ELIGIBILITY:
PATIENTS - Inclusion Criteria:-

* They are aged 55 or older
* They are multimorbid patients that suffer from two or more of the following four conditions in various disease combinations (two conditions set as the minimum threshold):-
* Diabetes type 2
* Renal Failure with eGFR/GFR 30 - 59 (measured or estimated glomerular filtration rate)
* Heart Failure in compliance with NYHA I-II (New York Heart Association classification of heart failure)
* Mild or moderate depression
* They still live and generally plan on living in their home (or in the community) for the 12-month trial duration.
* They or their informal caregiver pass the ICT Handling Self-Check (see Deliverable D10.4, Annex 8.3) (i.e. they have access to and some familiarity with the use of ICT).
* They, or their informal caregiver, have stable access to the internet and at least one of the following devices readily available to use the C3-Cloud components: Computer; Notebook; Smartphone; Tablet. This includes the use of Internet Browsers to open the C3-Cloud patient dashboards online.
* They are able to provide informed consent.

PATIENTS - Exclusion Criteria:-

•The exclusion criteria include almost completely the reverse of the inclusion criteria. Patients are not eligible for recruitment if:-

* They are aged 54 or below
* They suffer from any of the following conditions:
* Severe Renal Failure with eGFR/GFR <30
* Severe Heart Failure in compliance with NYHA III-IV
* Severe depression
* They have other debilitating conditions that impair their decision making capability or their life expectancy (e.g. end-of-life patients or cancer patients)
* They or their informal caregivers do not pass the ICT Handling Self-Check (i.e. they do not have access to suitable IT devices and do not have some familiarity with the use of ICT).
* They have disabilities or other health conditions that would prevent their active involvement in the study project or which prevent them from carrying out essential functions of the trial.
* They live in a care institution, for instance in a residential home or nursing home.
* Their health care expenses are covered by a private insurance: in the C3-Cloud pilot sites, private insurances have no data exchange with EHRs.
* They do not speak the regional language: English for SWFT; Spanish for the Basque country; Swedish for RJH
* They are unable to provide informed consent for study participation.

Patients with further chronic diseases and other co-morbidities or symptoms, for example, frailty, sleeping problems, malnourishment or anxiety, will not be excluded from recruitment. Informal caregivers who pass the ICT Handling Self-Check can substitute for the patient if the patient does not pass the ICT Handling Self-Check - the patient-informal caregiver pair can then still be recruited.

PATIENT'S HELPERS/CARERS - Exclusion Criteria:-

There are no specific inclusion criteria for informal caregivers. However, the following exclusion criteria apply:-

* They are aged 17 or below
* They do not have some familiarity with the use of ICT or do not have the capability to help the patient out with ICT usage if necessary.
* They do not have stable access to the internet and at least one of the following devices readily available to use the C3-Cloud components: Computer; Notebook; Smartphone; Tablet. This includes the use of Internet Browsers to open the C3-Cloud patient dashboards online.
* They are not available most of the time in person or via telephone, email, SMS or other means as to respond to calls for help.
* They have debilitating conditions that impair their decision-making capability.
* They do not speak the local language: English for SWFT; Spanish for the Basque country; Swedish for RJH

HEALTHCARE PROFESSIONALS - Inclusion Criteria:-

* normally be involved in the selected patients care
* open to new ways of working, specifically as part of a MDT (including GPs; consultant nurses or specialist nurses; district nurses; social workers; consultants; physiotherapists or pharmacists)
* open to the use of new technology: MDT members do not have to be technologically knowledgeable but they should be willing to learn how to use technology to support their work.

HEALTHCARE PROFESSIONALS - Exclusion Criteria:-

* None specific. Reverse of the above

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability & usefulness of the C3-Cloud system | 12 months
  This is qualitative research so the primary outcome measure will be the acceptability and usefulness of the technology by patients, informal care givers and health & care professionals. The UTAUT questionnaire (Unified Theory of Acceptance and User of Technology) will be performed to determine C3-Cloud user responses along the following UTAUT categories: performance expectancy, effort expectancy, social influence, cultural and language factors, technology anxiety, adoption timeline and associated facilitating conditions on the intended adoption behaviour. The questionnaire will be performed online and data will be aggregated completely anonymously using the online questionnaire platform "LimeSurvey", hosted on servers of empirica. The ordinal responses (e.g. "I strongly disagree" or "I strongly agree") are clustered along the UTAUT categories analsed anonymously.

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros N. Arvanitis, Study Chair — University of Warwick
Locations (3):
- Osakidetza, Vitoria-Gasteiz, Araba, Spain
- Region Jamtland Harjedalen, Östersund, Sweden
- South Warwickshire NHS Foundation Trust, Warwick, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only anonymised, aggregated data will be shared with researchers.

REFERENCES:
- [Derived] von Tottleben M, Grinyer K, Arfa A, Traore L, Verdoy D, Lim Choi Keung SN, Larranaga I, Jaulent MC, De Manuel Keenoy E, Lilja M, Beach M, Marguerie C, Yuksel M, Laleci Erturkmen GB, Klein GO, Lindman P, Mar J, Kalra D; C3-Cloud Research Team; Arvanitis TN. An Integrated Care Platform System (C3-Cloud) for Care Planning, Decision Support, and Empowerment of Patients With Multimorbidity: Protocol for a Technology Trial. JMIR Res Protoc. 2022 Jul 13;11(7):e21994. doi: 10.2196/21994. PMID 35830239
- See also: C3-Cloud Website — http://www.c3-cloud.eu/